CLINICAL TRIAL: NCT00006193
Title: Effectiveness of Atkins Diet for Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0761; M01RR000036 (NIH)
Record Dates: First submitted 2000-09-07; First posted 2000-09-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet

INTERVENTIONS:
Behavioral: diet

SUMMARY:
Dr. Atkins' New Diet Revolution has sold over 10 million copies and has been on the New York Times best seller list for 158 weeks. This and other low-carbohydrate diets, such as the ZONE, Sugar Busters, and the Carbohydrate Addicts Diet, have attracted much popular attention but little scientific evaluation. Given the widespread use of these diets, it seems prudent to evaluate them both for safety and efficacy. Therefore, the purpose of the study is to compare the effectiveness of two different weight control programs over the course of 52 weeks. These two programs are 1) the Atkins' New Diet Revolution, a low-carbohydrate, high-protein diet, and 2) Brownell's LEARN Program, a high carbohydrate, low fat diet based on behavior modification. Specifically, this study will compare short-term changes in weight, food intake, blood chemistries and mood in adult males (n=10) and females (n=10) who are randomized to either the Atkins' Diet or the LEARN Program for a period of one year. During this year, they will be under medical supervision. We will examine the effect of the two weight loss plans on changes in lipids, blood pressure, insulin sensitivity and ketones, and eating behavior. This is a feasibility study and thus the data will ultimately be used to design a large randomized trial with adequate statistical power.

ELIGIBILITY:
- BMI 25-40 kg/m2 inclusive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States